CLINICAL TRIAL: NCT00039156
Title: An Open Phase II Multi-Center Trial of BAY 59-8862 in Patients With Aggressive Refractory Non-Hodgkin's Lymphoma
Brief Title: BAY 59-8862 in Treating Patients With Refractory Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069358; THERADEX-100389; BAYER-100389; SUNY-HSC-4553
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2004-01

CONDITIONS: Lymphoma
Keywords: recurrent grade 3 follicular lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell | interventions — IDN 5109

INTERVENTIONS:
Drug: ortataxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BAY 59-8862 in treating patients who have refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall tumor response rate, including complete response (CR) and partial response (PR) rate, in patients with aggressive refractory non-Hodgkin's lymphoma treated with BAY 59-8862.
* Determine the overall survival in patients treated with this drug.
* Determine the time to progression in patients treated with this drug.
* Determine the duration of response (CR and PR) in patients treated with this drug.
* Determine the qualitative and quantitative toxicity profile of this drug in this patient population.
* Determine the pharmacokinetic profile of this drug in selected patients.

OUTLINE: This is a multicenter, open-label study.

Patients receive BAY 59-8862 IV over 1 hour on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months thereafter for up to 2 years.

PROJECTED ACCRUAL: A total of 20-140 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive refractory non-Hodgkin's lymphoma (NHL) of one of the following classifications, and for which chemotherapy is deemed appropriate:

  * Diffuse large B-cell lymphoma
  * Transformed NHL
  * Follicular large cell lymphoma
  * Peripheral T cell lymphoma
  * Anaplastic large cell lymphoma
  * Mantle cell lymphoma
  * Unclassified aggressive histology
  * Immunoblastic lymphoma
* Failed at least 1 prior therapy (primary resistant) OR
* Previously achieved a remission and then progressed or relapsed within 6 months of therapy
* At least 1 bidimensionally measurable lesion

  * Lesions within a previously irradiated field are not considered measurable
* No relapse within 6 months after prior autologous bone marrow transplantation
* No prior allogeneic bone marrow or stem cell transplantation or post-transplant lymphoproliferative disorder
* No parenchymal or meningeal CNS involvement unless the patient received prior definitive therapy more than 6 months ago, has had a negative imaging study within the past 4 weeks, and is clinically stable with respect to the tumor at study entry

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic:

* Total bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT and AST no greater than 2.0 times ULN (5.0 times ULN if hepatic involvement)
* PT, INR, and PTT less than 1.5 times ULN
* No chronic hepatitis B or C

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No clinically evident congestive heart failure
* No New York Heart Association class III or IV heart disease
* No serious cardiac arrhythmias
* No active coronary artery disease or ischemia

Other:

* No prior hypersensitivity to taxane compounds
* No known or suspected allergy to the investigational study agent or any agent given in association with this study
* No other prior or concurrent malignancy except basal cell skin cancer or curatively treated carcinoma in situ of the bladder or cervix (adequately cone biopsied)
* No substance abuse or medical, psychological, or social conditions that would preclude study participation
* No active clinically serious infections
* No other condition that is unstable or would preclude study participation
* No grade 2 or greater pre-existing peripheral neuropathy
* No history of seizure disorder

  * Prior seizures related to brain metastases allowed provided that the patient has been seizure-free for at least 2 months
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* See Chemotherapy
* At least 4 weeks since prior anticancer immunotherapy
* At least 3 weeks since prior biologic response modifiers (e.g., filgrastim [G-CSF])
* No concurrent anticancer immunotherapy
* No concurrent prophylactic G-CSF
* Concurrent G-CSF or other hematopoietic growth factors for acute toxicity (e.g., febrile neutropenia) allowed
* Concurrent chronic epoetin alfa allowed provided no dose adjustment occurred within 2 months prior to study

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior anticancer chemotherapy
* No more than 3 prior systemic chemotherapy regimens for metastatic NHL:

  * High-dose therapy for autologous hematopoietic stem cell transplantation (SCT) is considered 1 prior regimen
  * Salvage chemotherapy followed by autologous bone marrow transplant or peripheral SCT is considered 1 prior regimen
  * Antibody treatment is not considered 1 prior regimen
* No prior taxanes or oxaliplatin
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* Patients with prior parenchymal or meningeal CNS involvement:

  * No concurrent acute or tapered steroid therapy
  * Concurrent chronic steroid therapy allowed provided the dose is stable for 1 month before and after screening radiographic studies

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* Concurrent palliative radiotherapy allowed provided:

  * No progressive disease
  * No more than 10% of bone marrow is irradiated
  * Radiation field does not encompass a target lesion
* No other concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major surgery

Other:

* At least 4 weeks since prior investigational drugs
* No other concurrent investigational therapy or approved anticancer therapy
* No concurrent illicit drugs or other substances that would preclude study
* Concurrent therapeutic anticoagulants (e.g., warfarin or heparin) allowed provided there is no prior evidence of underlying abnormality with PT, INR, or PTT
* Concurrent nonconventional therapies (e.g., herbs or acupuncture) or vitamin/mineral supplements allowed provided that they do not interfere with study endpoints
* Concurrent bisphosphonates for prophylaxis or bone metastases allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: Rasim Ahmet Gucalp, MD, Study Chair — Montefiore Medical Center
Locations (15):
- United States (13):
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - HemOnCare, P.C., Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - West Clinic, Memphis, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - St. Paul's Hospital - Vancouver, Vancouver, British Columbia